CLINICAL TRIAL: NCT01304836
Title: Investigating New Onset Diabetes Mellitus in Kidney Transplant Recipients Receiving an Advagraf-Based Immunosuppressive Regimen With or Without Corticosteroids - A Multicenter, Two Arm, Randomized, Open Label Clinical Study
Brief Title: A Study Looking at Diabetes in Kidney Transplant Recipients Receiving Immunosuppressive Regimen With or Without Steroids
Acronym: ADVANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMR-EC-1211; 2010-019638-28 (EudraCT Number)
Record Dates: First submitted 2011-02-03; First posted 2011-02-28 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Kidney Transplantation
Keywords: Kidney; Diabetes Mellitus; Transplant; Immunosuppression
MeSH Terms: conditions — Diabetes Mellitus | interventions — Mycophenolic Acid; Basiliximab; Adrenal Cortex Hormones; Prednisolone; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10 Days of Steroids (Active Comparator): Advagraf + Basiliximab + MMF + Steroids (10 days)
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Simulect; Drug: Corticosteroids
- Optional Steroid bolus only (Experimental): Advagraf + Basiliximab + MMF + Steroids (bolus only)
  Interventions: Drug: Advagraf; Drug: Mycophenolate Mofetil; Drug: Simulect; Drug: Corticosteroids

INTERVENTIONS:
Drug: Advagraf — oral
  Other Names: FK506E; modified release tacrolimus
Drug: Mycophenolate Mofetil — oral
  Other Names: CellCept
Drug: Simulect — IV
  Other Names: Basiliximab
Drug: Corticosteroids — IV & oral
  Other Names: prednisolone; methylprednisolone

SUMMARY:
The purpose of this study is to focus on potential differences in the occurrence of new-onset Diabetes Mellitus (a glucose metabolism disorder) when two different regimens of immunosuppressive treatment are compared.

DETAILED DESCRIPTION:
The primary objective of this study is to compare an Immunosuppressive regimen with 10 days of corticosteroids with a regimen with only an optional intra-op bolus of corticosteroids with regard to incidence of new onset Diabetes Mellitus as per the American Diabetic Association (ADA) criteria at any point up to 24 weeks after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* End stage kidney disease and a suitable candidate for primary

kidney transplantation or re-transplantation (unless the graft was

lost from rejection within one year)

* Receiving a kidney transplant from a deceased or living (non

Human Leukocyte Antigen identical) donor with compatible AB0 blood type

* Female subjects of childbearing potential must have a

negative serum or urine pregnancy test at enrollment and must

agree to maintain highly effective birth control during the study.

A highly effective method of birth control is defined as those

which result in a low failure rate (CPMP/ICH/286/95 modified)

of less than 1% per year when used consistently and correctly

such as implants, injectables, combined oral contraceptives,

some IUDs, sexual abstinence or vasectomized partner

Exclusion Criteria:

* Receiving or having previously received an organ transplant

other than a kidney

* Cold ischemia time of the donor kidney > 30 hours
* Panel Reactive Antibody >20% (Highest level in 6 months prior to transplant)
* Previous renal transplant lost within one year for immunological reasons
* Receiving a graft from a non-heart-beating donor other than of Maastricht category 3 (withdrawal of support awaiting cardiac arrest)
* Significant liver disease, defined as having continuously

elevated SGPT/ALT and/or SGOT/AST and/or total bilirubin

levels ≥ 2 times the upper value of the normal range of the

investigational site or is receiving a graft from a hepatitis C or B

positive donor

* Diagnosis of Diabetes Mellitus prior to transplantation (treated with prescribed medications or diet controlled) or where there is evidence of a previous positive Oral Glucose Tolerance Test (OGTT) in the patients medical history or previous diagnosis of gestational diabetes or pre-baseline HbA1C ≥6.5%
* Requiring initial sequential or parallel therapy with immunosuppressive antibody preparation(s).
* Requiring ongoing dosing with a systemic immunosuppressive drug prior to transplantation (e.g. for Lupus Disease, FSGN etc) other than minimal levels of immunosuppressant following failure of a previous transplantation without nephrectomy
* Where Physician considers long term steroid treatment is necessary for the prevention of recurrent auto immune mediated renal disease or if the subject requires ongoing dosing with corticosteroids during the study for any other condition
* Significant, uncontrolled concomitant infections and/or severe diarrhea, vomiting, active upper gastro-intestinal tract malabsorption or active peptic ulcer
* Pregnant woman or breast-feeding mother
* Subject or donor known to be HIV positive
* Known allergy or intolerance to tacrolimus, macrolide antibiotics, corticosteroids, basiliximab, mycophenolate mofetil or any of the product excipients
* Evidence of malignant disease within the last 5 years other than Basal Cell Carcinoma or Squamous Cell Carcinoma
* Currently participating in another clinical trial and/or has taken an investigational drug within 28 days prior to randomization
* Any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator
* Unlikely to comply with the visits scheduled in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1166 (Actual)
Dates: Start 2011-01-22 (Actual); Primary Completion 2013-05-22 (Actual); Study Completion 2013-05-22 (Actual)

PRIMARY OUTCOMES:
Diagnosis of new onset Diabetes Mellitus as per ADA criteria at any point up to 24 weeks after kidney transplantation | up to 6 months

SECONDARY OUTCOMES:
Efficacy failure using a composite endpoint consisting of graft loss, biopsy confirmed acute rejection or graft dysfunction | up to 6 months
Positive Oral Glucose Tolerance Test | 8 weeks
Repeat Positive Oral Glucose Tolerance Test | 6 months
Renal function | at 6 months
Acute Rejections | up to 6 months
Biopsy confirmed acute rejections | up to 6 months
Subject survival | up to 6 months
Graft survival | up to 6 months
Change from Baseline in HbA1C levels | Baseline, week 12 and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe Ltd.
Locations (86):
- Australia (2):
  - Perth
  - Sydney
- Belgium (3):
  - Brussels
  - Leuven
  - Liège
- Cali, Colombia
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- Tartu, Estonia
- Helsinki, Finland
- France (12):
  - Bordeaux
  - Cité Nord
  - D'Angers
  - Le Puytren
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Rennes
  - Rouen
  - Strasbourg
  - Suresnes
- Germany (10):
  - Aachen
  - Bonn
  - Düsseldorf
  - Essen
  - Halle
  - Kaiserslautern
  - Mannheim
  - München
  - Regensburg
  - Rostock
- Hungary (2):
  - Debrecen
  - Szeged
- Italy (11):
  - Ancona
  - Bologna
  - Cagliari
  - L’Aquila
  - Milan
  - Padua
  - Pisa
  - Roma
  - Salerno
  - Treviso
  - Vicenza
- Riga, Latvia
- Vilnius, Lithuania
- Mexico (2):
  - Cuernavaca
  - Mexico City
- Maastricht, Netherlands
- Olso, Norway
- Poland (5):
  - Bydgoszcz
  - Gdansk
  - Poznan
  - Szczecin
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Romania (2):
  - Bucharest
  - Lasi
- Russia (6):
  - Moscow
  - Nizhny Novgorod
  - Omsk
  - Saint Petersburg
  - Vol’skiy
  - Yekaterinburg
- Slovakia (3):
  - Banská Bystrica
  - Bratislava
  - Košice
- Seoul, South Korea
- Spain (9):
  - Alicante
  - Barcelona
  - Córdoba
  - Madrid
  - Santa Cruz de Tenerife
  - Seville
  - Toledo
  - Valencia
  - Valladolid
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala
- Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Mourad G, Glyda M, Albano L, Viklicky O, Merville P, Tyden G, Mourad M, Lohmus A, Witzke O, Christiaans MHL, Brown MW, Undre N, Kazeem G, Kuypers DRJ; Advagraf-based immunosuppression regimen examining new onset diabetes mellitus in kidney transplant recipients (ADVANCE) study investigators. Incidence of Posttransplantation Diabetes Mellitus in De Novo Kidney Transplant Recipients Receiving Prolonged-Release Tacrolimus-Based Immunosuppression With 2 Different Corticosteroid Minimization Strategies: ADVANCE, A Randomized Controlled Trial. Transplantation. 2017 Aug;101(8):1924-1934. doi: 10.1097/TP.0000000000001453. PMID 27547871
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=212